CLINICAL TRIAL: NCT02564094
Title: Optimizing Treatment of the Anaemia in Onco-Hematological Diseases With NeoRecormon 30,000 IU Once Weekly
Brief Title: A Study of Epoetin Beta (NeoRecormon) in Participants With Solid Tumors or Hematologic Malignancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18043
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin beta (Experimental): Participants with hematologic or solid malignancies will receive epoetin beta for a treatment period of approximately 20 weeks.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Participants will receive SC epoetin beta as 30,000 international units (IU) once weekly for 20 weeks.
  Other Names: NeoRecormon

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacoeconomics of treatment with subcutaneous (SC) epoetin beta (NeoRecormon) in participants with hematologic malignancies or solid tumors. The anticipated time on study treatment is 20 weeks, and the target sample size is 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Multiple myeloma (MM), low-grade non-Hodgkin's lymphoma (NHL), chronic lymphocytic leukemia (CLL), breast cancer, lung cancer, or ovarian cancer
* Anemia with low erythropoeitin (EPO) levels

Exclusion Criteria:

* Poorly controlled hypertension
* Relevant acute or chronic bleeding requiring therapy within 3 months before study drug
* Treatment with EPO within the last 6 weeks
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate according to hemoglobin level | At Week 4
Transfusion requirement rate | From Weeks 5 to 12
Predictive value of reticulocyte increase | At Week 2

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (4):
- Bulgaria (4):
  - Plovdiv
  - Sofia
  - Stara Zagora
  - Varna